CLINICAL TRIAL: NCT07236385
Title: Artificial Intelligence Training Program Versus Standard Correction for Forward Head and Rounded Shoulder in Non-specific Neck Pain
Brief Title: AI Training Program vs Standard Correction for Forward Head and Rounded Shoulder in Neck Pain
Acronym: AI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, RANEEM MAHMOUD ELSHERIEF, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005976
Record Dates: First submitted 2025-09-13; First posted 2025-11-19 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Forward Head Posture; Rounded Shoulder Posture; Upper Cross Syndrome
Keywords: forward head and rounded shoulder posture ,hyperkyphosis OR "thoracic kyphosis
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI based exercise (Experimental): receive AI-generated personalized exercise regimens from the APECS-AI app
  Interventions: Other: AI based exercise
- standard corrective exercises (Active Comparator)
  Interventions: Other: standard corrective exercises

INTERVENTIONS:
Other: AI based exercise — receive AI-generated personalized exercise regimens from the APECS-AI app
  Arms: AI based exercise
Other: standard corrective exercises — Each exercise session begins with 10 min of warm-up activity and ends with 5 min of cool-down. Selected exercises will be designed in two phases: first, and second phases. Exercises will be progressed in frequency and intensity during these phases
  Arms: standard corrective exercises

SUMMARY:
this study will be to evaluate the effectiveness of AI-recommended exercise interventions versus standard corrective exercises in management of non-specific neck pain with forward head and rounded shoulder posture. with the goal of improving neck pain, functional disability, forward head, and rounded shoulder postures.

DETAILED DESCRIPTION:
The aim of the current study is to evaluate the efficacy of APECS-AI app suggested exercises and standard corrective exercises in managing non-specific neck pain with forward head and rounded shoulders posture. Forty-six subjects of both genders between (18 and 35 years old) have non-specific neck pain with forward head and rounded shoulder posture will be enrolled in this study. The subjects will be randomized into two equal groups (n = 23 each): An intervention group (Group A), will receive AI-generated personalized exercise regimens from the APECS-AI app, and a control group (Group B), will perform standard corrective exercises

ELIGIBILITY:
Inclusion Criteria: Subjects with non-specific neck pain who had localized neck pain felt it anywhere along the cervical spine, from the superior nuchal line to the first thoracic spinous process.

Neck pain between 3 and 8cm on a visual analogue scale. Subjects suffering from chronic (> 12 weeks) neck pain. Subjects with forward head posture with craniovertebral angle (CVA) angle less than 50 degrees.

Subjects with rounded shoulder posture as shoulder angle < 52. Subjects must not have received any pharmacological medication related to their musculoskeletal condition as non-steroidal anti-inflammatory drugs or muscle relaxant for at least three months prior to enrolment in the study.

Subjects must not have involved in any form of physical therapy or structured postural correction programs within the 6 months prior to study -

Exclusion Criteria:

1. Musculoskeletal diseases, cardiopulmonary diseases, and a history of surgery that could affect the experiment.
2. History of cervical spine injury or surgery.
3. Neck pain secondary to other conditions (e.g. Neoplasm, neurological diseases or vascular diseases).
4. Spondylosis and spondylolisthesis
5. A neurological disease, infection.
6. Inflammatory arthritis in the cervical spine.
7. Poor general health status that would interfere with the exercises -

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-11-30 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
The craniovertebral angle | 6 weeks
  forward head posture. will be measured by Kinovea software and the APECS AI app. More than 50 degrees is considered normal.
Shoulder angle | 6 weeks
  rounded shoulder posture will be measured by Kinovea software and the APECS AI app. more than 52 is considered normal
functional disability | 6 weeks
  is measured by neck disability index (NDI). A higher score reflects a greater level of neck disorder-related disability
pain level | 6 weeks
  It is measured by visual analogue scale (VAS). 10-cm line that represents a pain spectrum between "no pain" and "worst pain," as the word descriptions "no pain" on the left and "worst imaginable pain" on the right serve as anchors for the 100-mm-long horizontal line

CONTACTS AND LOCATIONS:
Overall Officials: NESREEN FAWZY MAHMOUD, Study Director — Lecturer of Physical Therapy for Musculoskeletal Disorders and Its Surgery Faculty of Physical Therapy Cairo University; PROF. Dr. ENAS FAWZY YOUSSF, Study Chair — Professor and Chairperson of Department of Physical Therapy for Musculoskeletal Disorders and Its Surgery Faculty of Physical Therapy Cairo University
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://download.cnet.com/apecs-ai-posture-evaluation-and-correction-system/3000-2129_4-78218468.html